CLINICAL TRIAL: NCT01764191
Title: [18 F]-Fluorodeoxyglucose (18F-FDG) Positron Emission Tomography (PET) in Cardiac Sarcoidosis
Brief Title: 18F-FDG PET Imaging in Cardiac Sarcoidosis
Status: Approved for marketing | Type: Expanded Access
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: BCCA-Cardiac PET
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — Fluorodeoxyglucose F18

INTERVENTIONS:
Other: 18F-Fluorodeoxyglucose (18F-FDG) PET/CT — All subjects suspected of cardiac sarcoidosis will receive an intravenous dose of 18F-FDG (determined by weight, but not to exceed 521 MBq). Following an uptake phase of about 60 minutes, each subject will receive a PET/CT scan to evaluate the presence of cardiac sarcoidosis.

SUMMARY:
This study has been designed to provide patients suspected of having cardiac sarcoidosis (CS) with a potentially diagnostic 18F FDG PET/CT. CS is difficult to diagnose with currently available methods, therefore this project will allow access to 18F FDG PET/CT scanning, which may more accurately diagnose the presence of CS. This study will also provide additional data to further examine the effectiveness and safety profile of 18F FDG for this condition. Accurate and early detection is important to allow for better management of CS and improve patient care.

The purpose of this study is to provide access to 18F-FDG PET/CT imaging in patients with clinical suspicion of cardiac sarcoidosis, and to collect additional data about the safety and effectiveness of 18F-FDG PET/CT in this patient population

DETAILED DESCRIPTION:
1. Purpose:The purpose of this study is to provide access to 18F-FDG PET/CT imaging in patients with clinical suspicion of cardiac sarcoidosis, and to collect additional data about the safety and effectiveness of 18F-FDG PET/CT in this patient population.
2. Hypothesis:18F-FDG PET/CT has greater sensitivity, specificity, and accuracy compared to the current clinical gold standard of diagnosis for CS, the Japanese Ministry of Health, Labour, and Welfare (MHLW) guidelines
3. Justification:Currently a clinical diagnosis CS is diagnosed using a combination of diagnostic techniques including imaging and biopsy. Biopsies are challenging as it can be difficult to locate the disease or access the desired biopsy location. MRI has been proven effective but it is limited as patients with pacemakers and cardioverter-defibrillators or patients with renal impairments are unable to have an MRI. Finally radionuclide scintigraphy with Gallium-67 or Thallium-201 (201Tl) has been useful, but can be non-specific for sarcoidosis. 18F-FDG PET/CT has significant advantages over other radionuclide imaging modalities due to superior resolution of PET coupled with the affinity of inflammatory cardiac tissue to metabolize FDG. 18F-FDG PET/CT has been found to have higher sensitivity and specificity over other conventionally used imaging modalities.
4. Research Method:This will be an expanded access study in which adult subjects with a clinical suspicion of CS will be invited to participate, in order to identify potential sites for biopsy or provide confirmation of the presence of CS. Based on population extrapolation from all diagnosed or suspected cases of CS in British Columbia (BC), as well as expert clinical opinion, it is estimated that 10 to 15 patients per year will be enrolled in the study. Over a three year period, the expected sample size will be 30 - 45 patients. All subjects will receive an 18F-FDG PET/CT at the BC Cancer Agency (BCCA) - Vancouver Centre.
5. Statistical Analysis:The planned sample size is 150 patients. The primary endpoint is to provide PET/CT imaging to patients diagnosed with or suspected of CS. The secondary end-point will be to assess the sensitivity, specificity and accuracy of 18F-FDG PET in BC population. Confidence intervals of 95% will be used to assess this using exact binomial distribution. All analyses will be performed in direct consultation with a qualified statistician.

Sensitivity (ratio of true positive lesions to total positive lesions), specificity (ratio of true negative lesions to total negative lesions) and accuracy (ratio of total correct studies to the total number of biopsied lesions) of 18F-FDG PET studies performed by the BCCA will be obtained by comparing results of the PET scan with a composite of the outcome of clinical examinations, histopathological diagnosis, if those results are available, and results of all other available imaging (cardiac MRI, 201Tl, 67Ga). Confidence intervals (95% CI) for sensitivity, specificity and accuracy will be calculated using exact binomial distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 - 3.
* Able to provide written informed consent.
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 45 minutes and tolerating intravenous cannulation for injection.
* Clinical suspicion of cardiac sarcoidosis, including a combination of:

  * Patients with systemic sarcoidosis and symptoms suggestive of heart failure (eg. fatigue, dyspnea, edema etc.)
  * Idiopathic heart failure, particularly of preserved systolic function variety
  * Presentation with arrhythmia (eg. heart block, ventricular tachycardia, etc.)
  * Progressive heart failure symptoms not responding to conventional therapy
  * Other clinical presentations where in the experience of treating cardiologist cardiac sarcoid needs to be ruled out (ie. Heart transplant or ventricular assist device candidacy)
* Routine tests for CS are inconclusive, such as:

  * ECG
  * Holter
  * echocardiogram
  * 67Ga scintigraphy is inconclusive
  * Cardiac MRI is inconclusive or not possible to conduct
* Patient has renal dysfunction which limits other radionuclide imaging.

Exclusion Criteria:

* Patients blood glucose > 11.1 mmol/L (200 mg/dL) measured by glucometer immediately prior to scan.
* Patients with confirmed diabetes.
* Patients unable to comply with the dietary modifications or prolonged fasting as per trial protocol.
* Pregnancy.
* Patients who are medically unstable eg. acute cardiac or respiratory distress, or hypotensive.
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT machine (diameter 70 cm).

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada